CLINICAL TRIAL: NCT03931187
Title: Double ABCX Theory Based Cognitive Psychotherapy Combined Progressive Muscle Relaxation Intervention on Women Undergoing In Vitro Fertilization-Embryo Transfer Treatment
Brief Title: Double ABCX Theory Based Cognitive Psychotherapy Combined Progressive Muscle Relaxation Intervention on Women Undergoing IVF-ET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Anni Wang, Principal Investigator, Central South University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Intervention on IVF-ET
Record Dates: First submitted 2019-04-23; First posted 2019-04-30 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-11

CONDITIONS: Infertility
Keywords: cognitive psychotherapy; progressive muscular relaxation; in vitro fertilization and embryo transfer(IVF-ET); Couples Therapy
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Women intervention arm (Experimental): Intervention will be applied to the women within the couple.
  Interventions: Behavioral: Cognitive progressive muscular relaxation therapy
- Couple intervention arm (Experimental): Intervention will be applied to the couple, both men and women.
  Interventions: Behavioral: Cognitive progressive muscular relaxation therapy
- Control arm (No Intervention): The couple will receive the normal nursing care.

INTERVENTIONS:
Behavioral: Cognitive progressive muscular relaxation therapy — This therapy combines cognitive psychotherapy and progressive muscular relaxation, intervened 6 times with 1-1.5 hour each time. The whole therapy will last round 28-30 days during IVF-ET.
  Arms: Couple intervention arm; Women intervention arm

SUMMARY:
The in vitro fertilization and embryo transfer(IVF-ET) is a therapy to help the infertile couples. The mental health status of couple under IVF-ET, commonly seen in depression and anxiety, is found to be closely related to the success of IVF-ET. This study aims to develop a intervention program combing cognitive psychotherapy and progressive muscle relaxation to ease the negative emotion and promote the success rate among couples undergoing IVF-ET.

ELIGIBILITY:
Inclusion Criteria:

* The couple who are eligible for in vitro fertilization-embryo transfer (IVF-ET) treatment;
* Junior high school and above;
* voluntarily accepted for investigation and signed informed consent.

Exclusion Criteria:

* Suffering from physical diseases such as severe heart, liver and kidney, and mental disorders;
* Experiencing major traumatic events in the past 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological sex
Enrollment: 67 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Change of depression score | The investigators will measure the socre of depression at baseline and immediately after intervention ( the duration of intervention is around 1 month).
  The Self-reported Depression Scale （SDS）will be used to assess the score of depression.The total score of SDS ranges from 0-80, with 40 as the cutoff. The higher the total score, the more depressive.
Change of anxiety score | The investigators will measure the socre of anxiety at baseline and immediately after intervention ( the duration of intervention is around 1 month).
  The Self-reported Anxiety Scale (SAS) will be used to assess the score of anxiety.The total score of SAS ranges from 0-80, with 30 as the cutoff. The higher the total score, the more anxious.

SECONDARY OUTCOMES:
Change of Blood Cortisol | The investigators will measure the socre of Blood Cortisol at baseline and immediately after intervention ( the duration of intervention is around 1 month).
  This is a kind of hormone closely related to stress, and the investigators will measure the level of Blood Cortisol by Blood test.
Change of sleeping quality | The investigators will measure the socre of sleeping quality at baseline and immediately after intervention ( the duration of intervention is around 1 month).
  The physical condition closely related to stress. The investigators will use Self-Rating Scale of Sleep to measure the sleeping quality of the participants. The total sore ranges from 5 to 50, with higher score reflects better sleep quality.
Successful conception rate (%) | The doctor will test whether it is successfully conceived 4 weeks after the embryo is implanted. The last intervention is on the day of embryo implantation. The investigators will count this 4 weeks after completion of intervention.
  The investigators will count the successful conception rate at each arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Infertility Reproductive Center, Second Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
The participants are not willing to share the data.

REFERENCES:
- [Derived] Wang A, Zhang W, Li H, Guo Y, Yu NX, Zhang J. An 8-week community-based resilience group intervention for Chinese parents who lost their only child: A two-armed pragmatic waitlist-control trial. Psychol Trauma. 2025 Jan;17(1):225-234. doi: 10.1037/tra0001670. Epub 2024 Apr 22. PMID 38647487
- [Derived] Chen D, Wang A, Zhang W, Guo Y, Yao S, Chen X, Zhang J. Effectiveness of double ABCX-based psychotherapy for psychological distress among women undergoing in vitro fertilization-embryo transfer: a three-arm randomized controlled trial. J Psychosom Obstet Gynaecol. 2023 Dec;44(1):2278015. doi: 10.1080/0167482X.2023.2278015. Epub 2023 Dec 6. PMID 38056467

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT03931187/Prot_SAP_000.pdf